CLINICAL TRIAL: NCT03517514
Title: Investigating All-Cause 30-Day Hospital Readmisisons in Patients Discharged From a Tertiary Teaching Hospital With Acute Decompensated Heart Failure Diagnosis
Brief Title: Heart Failure Hospital Readmissions and Physical Therapy
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Bobby Belarmino PT,DPT,MA, Senior Physical Therapist (Level IV), The Methodist Hospital Research Institute
Other Study IDs: Pro00018201
Record Dates: First submitted 2018-04-06; First posted 2018-05-07 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Acute Heart Failure
Keywords: Heart Failure; Physical Therapy; Hospital Readmission
MeSH Terms: conditions — Heart Failure | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical Therapy service — routine physical therapy care

SUMMARY:
This is a dissertation study which is divided into three different studies in order to answer the main research question (Study 3). The primary aim of this research (dissertation) is to investigate all-cause 30-day hospital readmission using functional mobility (5mWT, 30STS, 6MWT, TUG), psychosocial attributes (KCCQ-12, HADS, ESSI), adherence to home exercise program, participation in a supervised exercise program, and number of follow up checkups with physicians or advanced health providers of patients with Acute Decompensated Heart Failure (ADHF) diagnosis who were discharged from a tertiary teaching hospital.

Study 1: What is the effect of acute physical therapy on functional ability in individuals admitted with ADHF? Study 2: What is the effect of acute physical therapy on psychosocial attributes in individuals admitted with ADHF? Study 3: Which factors such as functional mobility (5mWT, 30STS, 6MWT, TUG), psychosocial attributes (KCCQ-12, HADS, ESSI), adherence to home exercise program, participation in a supervised exercise program, and number of follow up checkups with physicians or advanced health providers predict all-cause 30-day hospital readmission in patients discharged from a tertiary, teaching hospital with ADHF diagnosis?

DETAILED DESCRIPTION:
The research plan is to investigate how acute physical therapy can play a big role in lowering 30-day hospital readmission in patients discharged with acute decompensated heart failure (ADHF). Several factors will be used to investigate and predict 30-day hospital readmission. Such factors are (1) functional mobility; 2) psychosocial attributes; (3) number of follow ups with providers; (4) adherence to home exercise program; (5) and participation in a supervised exercise program. Functional mobility will be measured by four different functional outcome measurements such as 5 meter walk test (5mWT), 30 seconds sit to stand test (30STS), six minute walk test (6MWT), and time up and go test (TUG). The psychosocial attributes will be measured by three different, pen and paper, self-survey questionnaires namely Kansas City Cardiomyopathy Questionnaire-12 (KCCQ12), Hospital Anxiety and Depression Scale (HADS), ENRICHD Social Support Instrument (ESSI). Moreover, once the patient returns home, two phone surveys will be conducted (every two weeks) for a period of 30 days of hospital discharge as a follow up.

For the outcome measurements, the 5mWT is a simple test to measure individual's gait (walking) speed. The 30STS is a simple and easy test to complete in assessing functional lower extremity strength. The 30STS asks individual to stand up (assuming erect posture as much as possible with or without hands support) as many as possible from a regular chair with arm rest within 30 seconds timeframe. The 6MWT is simple and practical test is to measure aerobic capacity by measuring distance of an individual's ability to walk for 6 minutes. The TUG is to measure the time in seconds for a person to rise from sitting from a standard arm chair, rise, walk 10 feet, walk back to the previous arm chair, and sit down. The objective of the TUG test is to classify patient's fall risk. In addition, the functional mobility, basing on the functional outcome measures conducted, will be further assessed at the end of physical therapy service at the hospital by using Global Rating of Scale (GROC). The GROC is a self-survey using 5 point Likert scale, measuring how patient perceives the overall degree of change of improvement or perhaps a lack of improvement.

For the Psychosocial Measures, the Kansas City Cardiomyopathy Questionnaire (KCCQ)-12 is a shorter version of the original KCCQ tool. The objective of this test is to quantify self-measurement of physical function, symptoms, social function, self-efficacy and knowledge, and quality of life as it relates to their own heart failure diagnosis. The Hospital Anxiety and Depression Scale (HADS) is a self-reported questionnaire designed to measure the levels of anxiety and depression that an individual is experiencing. The objective of this tool is to serve as a screening tool to identify individuals who may suffer from anxiety and depression. The ENRICHD Social Support Instrument (ESSI) is a seven-item self-report survey that assesses patient's belief of their social support attributes (emotional, instrumental, informational, and appraisal).

ELIGIBILITY:
Inclusion Criteria:

* all admitted at Houston Methodist Hospital with a primary diagnosis of acute heart failure or similar type of medical diagnosis
* stable medical state (HR equal or greater than 50 bpm, mean BP of 60 mmHg or better, Oxygen saturation (with or without oxygen supplement) of 90% or better; RR of 15 or better
* 50 years old and over and able to follow 2 simple commands
* establish discharge recommendation to home settings
* ambulatory with or without assitive device(s)

Exclusion Criteria:

* history of psychiatric disorder
* diagnosis of acute kidney injury requiring continuous renal replacement therapy
* diagnosis of major cognitive impairment (dementia, Alzheimer's dse, etc)
* inability to read and understand basic english language
* establish discharge recommendation to post-acute care settings (e.g. SNF, inpatient rehab, LTACH)
* inability to complete any functional mobility test due to musculoskeletal or other disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All medically stable, admitted patients at the hospital that have an admitting diagnosis of acute heart failure (or similar diagnosis) will be screened as potential study participants.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
hospital readmission within 30 days | less than or equal to 30 days
  Identification of patient hospital readmission within 30 days of discharge (day 0).

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  Compare measured total walking distance (in feet) within 6 minutes time
30 seconds Sit to Stand Test (30STS) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  Measurement of the total number of times a patient can complete a sit to stand task within 30 seconds, using a standard chair with arm rest (quantity of tasks)
Five Meter Walk Test (5mWT) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  Measurement of walking speed (in meter/seconds) over a 5 meter walking distance
Time Up and Go Test of Fall Risk (TUG) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  To classify patient's risk of falls will measure the time (in seconds) it takes to complete the task of standing up from a chair, walk 10 feet, turn around, and return to previous sitting position.
Global Rating of Change Scale (GROC) | End of study (post-physical therapy; defined as time frame: Day 2 to 8 weeks)
  To rate a 4 question, 11 point Likert scale per question, regarding a person's perception of the change in (1) walking distance, (2) walking speed, (3) risk of falls, and (4) number of times of complete sit to stand task after completing acute physical therapy services

OTHER OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  A 23-item, self-administered subjective questionnaire, to measure the quality of life of individuals living with heart failure regarding their physical function, heart failure symptoms, social and physical function with a score of 0 to 100, where the higher the number, the better the health status.
Hospital Anxiety and Depresssion Scale (HADS) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  A self-reported score measuring the level of anxiety and depression in the past week where the total score of anxiety and depression is 0 to 21, with the higher range from 8- 21 as borderline to abnormal.
Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Social Support Instrument (ESSI) | Comparing any change between pre-physical therapy treatment (Day 1) to post-physical therapy treatment (defined as time frame: Day 2 to 8 weeks)
  Seven item self-reported survey to measure an individual's perceived level of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Bobby C Belarmino, PT,DPT,MA, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross JS, Chen J, Lin Z, Bueno H, Curtis JP, Keenan PS, Normand SL, Schreiner G, Spertus JA, Vidan MT, Wang Y, Wang Y, Krumholz HM. Recent national trends in readmission rates after heart failure hospitalization. Circ Heart Fail. 2010 Jan;3(1):97-103. doi: 10.1161/CIRCHEARTFAILURE.109.885210. Epub 2009 Nov 10. PMID 19903931
- [Background] Hernandez AF, Greiner MA, Fonarow GC, Hammill BG, Heidenreich PA, Yancy CW, Peterson ED, Curtis LH. Relationship between early physician follow-up and 30-day readmission among Medicare beneficiaries hospitalized for heart failure. JAMA. 2010 May 5;303(17):1716-22. doi: 10.1001/jama.2010.533. PMID 20442387
- [Background] Hines AL, Barrett ML, Jiang HJ, Steiner CA. Conditions With the Largest Number of Adult Hospital Readmissions by Payer, 2011. 2014 Apr. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #172. Available from http://www.ncbi.nlm.nih.gov/books/NBK206781/ PMID 24901179
- [Background] McIlvennan CK, Eapen ZJ, Allen LA. Hospital readmissions reduction program. Circulation. 2015 May 19;131(20):1796-803. doi: 10.1161/CIRCULATIONAHA.114.010270. No abstract available. PMID 25986448
- [Background] Yamada S, Shimizu Y, Suzuki M, Izumi T; PTMaTCH collaborators. Functional limitations predict the risk of rehospitalization among patients with chronic heart failure. Circ J. 2012;76(7):1654-61. doi: 10.1253/circj.cj-11-1178. Epub 2012 Apr 7. PMID 22484978
- [Background] Desai AS, Stevenson LW. Rehospitalization for heart failure: predict or prevent? Circulation. 2012 Jul 24;126(4):501-6. doi: 10.1161/CIRCULATIONAHA.112.125435. No abstract available. PMID 22825412
- [Background] McCabe N, Butler J, Dunbar SB, Higgins M, Reilly C. Six-minute walk distance predicts 30-day readmission after acute heart failure hospitalization. Heart Lung. 2017 Jul-Aug;46(4):287-292. doi: 10.1016/j.hrtlng.2017.04.001. Epub 2017 May 24. PMID 28551310
- [Background] DiDomenico RJ, Park HY, Southworth MR, Eyrich HM, Lewis RK, Finley JM, Schumock GT. Guidelines for acute decompensated heart failure treatment. Ann Pharmacother. 2004 Apr;38(4):649-60. doi: 10.1345/aph.1D481. Epub 2004 Feb 24. PMID 14982975
- [Background] Alhurani AS, Dekker RL, Abed MA, Khalil A, Al Zaghal MH, Lee KS, Mudd-Martin G, Biddle MJ, Lennie TA, Moser DK. The association of co-morbid symptoms of depression and anxiety with all-cause mortality and cardiac rehospitalization in patients with heart failure. Psychosomatics. 2015 Jul-Aug;56(4):371-80. doi: 10.1016/j.psym.2014.05.022. Epub 2014 Jun 2. PMID 25556571
- [Background] Fisher SR, Kuo YF, Sharma G, Raji MA, Kumar A, Goodwin JS, Ostir GV, Ottenbacher KJ. Mobility after hospital discharge as a marker for 30-day readmission. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):805-10. doi: 10.1093/gerona/gls252. Epub 2012 Dec 19. PMID 23254776
- [Background] Fisher SR, Graham JE, Ottenbacher KJ, Deer R, Ostir GV. Inpatient Walking Activity to Predict Readmission in Older Adults. Arch Phys Med Rehabil. 2016 Sep;97(9 Suppl):S226-31. doi: 10.1016/j.apmr.2015.09.029. Epub 2016 Jun 2. PMID 27264549
- [Background] Reeves GR, Whellan DJ, Duncan P, O'Connor CM, Pastva AM, Eggebeen JD, Hewston LA, Morgan TM, Reed SD, Rejeski WJ, Mentz RJ, Rosenberg PB, Kitzman DW; REHAB-HF Trial Investigators. Rehabilitation Therapy in Older Acute Heart Failure Patients (REHAB-HF) trial: Design and rationale. Am Heart J. 2017 Mar;185:130-139. doi: 10.1016/j.ahj.2016.12.012. Epub 2016 Dec 28. PMID 28267466
- [Background] Wilson CM, Kostsuca SR, Boura JA. Utilization of a 5-Meter Walk Test in Evaluating Self-selected Gait Speed during Preoperative Screening of Patients Scheduled for Cardiac Surgery. Cardiopulm Phys Ther J. 2013 Sep;24(3):36-43. PMID 23997690
- [Background] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Background] Tabata M, Shimizu R, Kamekawa D, Kato M, Kamiya K, Akiyama A, Kamada Y, Tanaka S, Noda C, Masuda T. Six-minute walk distance is an independent predictor of hospital readmission in patients with chronic heart failure. Int Heart J. 2014;55(4):331-6. doi: 10.1536/ihj.13-224. Epub 2014 Jun 5. PMID 24898596
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Herman T, Giladi N, Hausdorff JM. Properties of the 'timed up and go' test: more than meets the eye. Gerontology. 2011;57(3):203-10. doi: 10.1159/000314963. Epub 2010 May 20. PMID 20484884
- [Background] Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. Circ Cardiovasc Qual Outcomes. 2015 Sep;8(5):469-76. doi: 10.1161/CIRCOUTCOMES.115.001958. PMID 26307129
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Stern AF. The hospital anxiety and depression scale. Occup Med (Lond). 2014 Jul;64(5):393-4. doi: 10.1093/occmed/kqu024. No abstract available. PMID 25005549
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Vaglio J Jr, Conard M, Poston WS, O'Keefe J, Haddock CK, House J, Spertus JA. Testing the performance of the ENRICHD Social Support Instrument in cardiac patients. Health Qual Life Outcomes. 2004 May 13;2:24. doi: 10.1186/1477-7525-2-24. PMID 15142277
- [Background] Mitchell PH, Powell L, Blumenthal J, Norten J, Ironson G, Pitula CR, Froelicher ES, Czajkowski S, Youngblood M, Huber M, Berkman LF. A short social support measure for patients recovering from myocardial infarction: the ENRICHD Social Support Inventory. J Cardiopulm Rehabil. 2003 Nov-Dec;23(6):398-403. doi: 10.1097/00008483-200311000-00001. No abstract available. PMID 14646785
- [Background] Garrison C, Cook C. Clinimetrics corner: the Global Rating of Change Score (GRoC) poorly correlates with functional measures and is not temporally stable. J Man Manip Ther. 2012 Nov;20(4):178-81. doi: 10.1179/1066981712Z.00000000022. PMID 24179325
- [Background] Schmitt J, Abbott JH. Global ratings of change do not accurately reflect functional change over time in clinical practice. J Orthop Sports Phys Ther. 2015 Feb;45(2):106-11, D1-3. doi: 10.2519/jospt.2015.5247. Epub 2015 Jan 8. PMID 25573006
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Walenkamp MM, de Muinck Keizer RJ, Goslings JC, Vos LM, Rosenwasser MP, Schep NW. The Minimum Clinically Important Difference of the Patient-rated Wrist Evaluation Score for Patients With Distal Radius Fractures. Clin Orthop Relat Res. 2015 Oct;473(10):3235-41. doi: 10.1007/s11999-015-4376-9. Epub 2015 Jun 4. PMID 26040969
- See also: Heart Failure matters — http://www.heartfailurematters.org/en_GB
- See also: What is Heart failure? — http://www.heart.org/HEARTORG/Conditions/HeartFailure/AboutHeartFailure/About-Heart-Failure_UCM_002044_Article.jsp#.WtKHJMuWxUQ